CLINICAL TRIAL: NCT01229787
Title: The Relation Between Obesity, Adipose Tissue Content of Fatty Acids and Systemic and Airway Inflammation
Status: Completed | Type: Observational
Sponsor: Cyprus International Institute for Environment and Public Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr Panayiotis Yiallouros, Cyprus International Institute for the Environment and Public Health
Other Study IDs: CIIRespiratory1
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2009-07

CONDITIONS: Asthma, Allergies and Obesity
Keywords: asthma; allergies; obesity
MeSH Terms: conditions — Asthma; Hypersensitivity; Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Obesity has been recognized as a risk factors for developing asthma. In a cohort of 5384 children aged 15-17, we aim to:

1. To investigate the association of asthma prevalence at age 15-17 with body mass index (BMI) at age 15-17 and BMI at age 11-12 years Part II
2. To investigate the association of BMI in adolescence and BMI at age 11-12 years with:

   1. Prevalence of allergic sensitization
   2. Lung function
   3. Levels of airway inflammation at age 16-18 years
   4. Severity of asthma

Secondly, to assess diet and physical activity involvement as effect modifiers in these possible associations.

DETAILED DESCRIPTION:
Cross-sectional studies in Northern America, Northern Europe and Asia indicate an increased prevalence and severity of asthma in the obese whereas longitudinal studies have indicated that increasing BMI is associated with increased risk of incident asthma in women. However, the mechanisms through which where-by obesity increases the risk for asthma remain unclear. There are only few studies from North America and Asia that suggested that obesity is associated with increased skin test reactivity and atopic diseases and many more that suggest obesity has no association with atopy. In adult asthmatics, it has also been shown that both medical and surgical weight loss is consistently associated with dramatic improvements in lung function, asthma symptoms, and medication usage. However, in children no study has elaborated on the potential benefits of reducing weight.

Total fat intake has also been associated with the diagnosis of asthma. N-3 fatty acids have been noted to inversely correlate with body fat, while levels of N-6 fatty acids correlated positively with body fat. Increased dietary intake of N-3 fatty acid (such as eicosapentaenoic acid) (mainly fish oils) has been generally associated with protection from asthma, while intake of N-6 fatty acids (such as linoleic acid) may increase asthma risk, although this remains controversial. Linoleic acid may act as a precursor of arachidonic acid which subsequently serves as a precursor of 4-series leukotrienes that are highly active mediators of inflammation.

There are only two studies that investigated the levels of exhaled nitric oxide (ENO) as indicator of airway inflammation in relation with obesity and asthma. One study showed significant increase of ENO with increasing BMI in healthy adults. However, the levels of ENO and exhaled leukotriene B4 were recently found to be increased in lean and obese asthmatic children but not related to their BMI's.

In Southern European countries, there are no representative epidemiological data on the contribution of obesity to asthma burden. In this area of the world, there are also no studies on the effect of important lifestyle factors including diet and physical activity on the association of adiposity with asthma pathophysiology. In addition, no information exists on levels of airways inflammation both in non-asthmatics and asthmatics subjects in relation to body content in fat and the impact of weight reduction on airway inflammation.

In years 2001-2003, a national health survey was conducted in Cyprus focusing on nutrition and physical fitness of all children aged 11-12 years (attending the 6th form of all primary schools). With this project we proposed to approach this group of children in years 2007-2009 to investigate the following hypotheses:

AIMS:

The aims of the study are as follows:

Part I To investigate the association of asthma prevalence at age 15-17 with body mass index (BMI) at age 15-17 and independently with BMI at age 11-12 years Part II

To investigate the association of BMI at age 16-18 and independently of BMI at age 11-12 years with:

1. Prevalence of allergic sensitization
2. Lung function
3. Levels of airway inflammation at age 16-18 years
4. Severity of asthma

Secondly, to assess diet and physical activity involvement as effect modifiers in these possible associations.

PART I METHODOLOGY:

Study population Part I took place during the months of January 2007 to June 2007 and children attending the 1st (15-16 years) and 2nd (16-17 years) classes in all public and private Lyceia schools across the Republic of Cyprus were invited to participate. The targeted population were 19849 children that participated in an earlier study in years 2001-3 and had amongst other assessments anthropometric measurements, assessment of cardio-respiratory fitness and serum lipids taken at that time.

For the assessment of children's asthma status we used the Greek version of the ISAAC (International Study of Asthma and Allergies in Childhood) core questionnaire supplemented with questions relating to potential person-based risk factors such as the place of birth of the child, ethnic origin of the parents, birth order, parental education level, parental smoking, history of atopy in the immediate family (siblings and parents with a history of asthma, eczema and or hay fever), personal uptake of smoking, pet ownership and place of residence.

All participating students had also their weight, percentage body fat and Body Mass Index (BMI) measured. The subjects' BMI had been classified as normal weight, overweight or obese according to sex and age specific cut-offs (six months intervals), suggested by the International Obesity Task Force (IOTF).

Compilation of Dataset

An effort to match subjects on the 2007 cross-sectional database with subjects on the 2001-2002 old cross-sectional database was carried out using various matching parameters. A dataset of 5384 subjects was constructed with matched BMI values in 2007 (aged 15-17 years) and in 2001-2003 (aged 11-12 years).

Statistical Analysis

Using answers to the basic questions for asthma and respiratory morbidity of the ISAAC questionnaire the case definition was further refined to:

1. Active asthma: positive answers to questions on ever having asthma and current wheeze and or night time cough unrelated to colds in the past 12 months
2. Inactive asthma: positive answer to question on ever having asthma and negative answers to questions for current wheeze and night time cough unrelated to colds in the past 12 months
3. Respiratory symptoms without asthma: negative answer to question on ever having asthma and positive answer(s) to questions on current wheeze and or night time cough unrelated to colds in the past 12 months.

The associations between disease outcomes and obesity predictors (BMI z-score and body fat %), were analyzed through univariate analysis and the odds ratio (OR) were calculated with 95% confidence intervals (CI). In addition to the univariate analysis, multiple logistic regression was also performed to further investigate the associations of obesity predictors and disease outcomes adjusting for confounders and stratifying by significant effect modifiers. Statistical significance was set at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* not applicable

Exclusion Criteria:

* not applicable

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Part I took place in 2007 and children 15-16 and 16-17 years across Cyprus were invited to participate. The targeted population were 19849 children that participated in an earlier study in years 2001-3 and had anthropometric measurements, assessment of cardio-respiratory fitness and serum lipids taken at that time. The subjects of the second part of the study were selected from the 5384 subjects that had participated in the first part and had matched data on current and past BMI. We targeted subjects for part two of the study with the following criteria:1. Current Wheezers: All active asthmatics across all BMI subgroups. Definition of Current Wheezer: Positive answer to the question in ISAAC questionnaire: "Have you had wheezing in the past 12 months?" 2. Never Wheezers: 700 controls selected in a random way across all BMI groups. Definition of Never Wheezer: Negative answers to both of the following two questions: "Have you ever had wheezing?" and "Have you ever had asthma?"
Sampling Method: Non-Probability Sample
Enrollment: 5384 (Actual)
Dates: Start 2007-01; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The association between asthma prevalence in adolescence and obsity in adolescence and in childhood
  To investigate the association of asthma prevalence at age 15-17 with body mass index (BMI) at age 15-17 and at age 11-12 years

SECONDARY OUTCOMES:
Association of BMI in adolescence and in childhood with allergic sensitization and lung function
  To investigate the association of BMI in adolescence and BMI at age 11-12 years with:
  1. Prevalence of allergic sensitization
  2. Lung function
  3. Levels of airway inflammation at age 16-18 years
  4. Severity of asthma

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Yiallouros, MD, PhD, Principal Investigator — Cyprus International Insitute
Locations (1):
- Cyprus International insitute, Nicosia, Nicosia, Cyprus